CLINICAL TRIAL: NCT05501431
Title: Personalized Parkinson Project PSP Cohort
Acronym: PPP-PSP
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: UCB Pharma (Industry); Verily Life Sciences LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: NL75356.091.20
Record Dates: First submitted 2022-08-11; First posted 2022-08-15 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2024-09

CONDITIONS: Progressive Supranuclear Palsy; Brain Diseases; Neurodegenerative Diseases; Movement Disorders
Keywords: Progressive Supranuclear Palsy; Biomarkers; Wearable sensors; Disease progression
MeSH Terms: conditions — Supranuclear Palsy, Progressive; Brain Diseases; Neurodegenerative Diseases; Movement Disorders; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood specimen from all enrolled participants
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Progressive Supranuclear Palsy (PSP): Participants with possible or probable PSP, wearing the Verily Study Watch for 1 year.
  Interventions: Device: Verily Study Watch
- Healthy Controls (HC): Participants without a neurological condition, age and gender matched to the PSP cohort, , wearing the Verily Study Watch for 1 year.
  Interventions: Device: Verily Study Watch

INTERVENTIONS:
Device: Verily Study Watch — The Verily Study Watch is a smartwatch, collecting physiological and/or environmental information. The sensors collect data that include movement and activity, pulse rate, skin impedance, electrocardiogram (ECG), environmental temperature, and ambient light level.

SUMMARY:
There is an urgent need for the development of digital progression biomarkers, which are sensitive to detect small, but potentially clinically relevant changes in the disease course. Digital biomarkers are based on (i) continuously collected real-time data, during the patient's day to day activities; and (ii) task-based assessment. In this study the investigators are interested in developing algorithms for the detection of disease progression in PSP patients in key clinical parameters: bradykinesia, gait, rising from a chair and falls, based on (i) sensor data obtained by means of passive monitoring during daily living; and (ii) sensor data collected during the Virtual Motor Exam.

DETAILED DESCRIPTION:
Rationale In light of the advent of a wide range of new disease modifying treatments, and acknowledging that existing clinical outcome measures may well be insufficiently sensitive to detecting small but potentially clinically relevant changes in the disease course, there is an urgent need for development of digital progression biomarkers, not only in the field of Parkinson's disease, but also in the field of the various forms of atypical parkinsonism, including Progressive Supranuclear Palsy (PSP).

Study Design Prospective, longitudinal, single-center cohort study.

Study Objectives The primary objective is to develop algorithms for the detection of disease progression in PSP patients in key clinical parameters: bradykinesia, gait, rising from a chair and falls, based on (1) sensor data obtained by means of passive monitoring during daily living; and (2) sensor data collected during the Virtual Motor Exam.

The second objective of this study is to create a longitudinal dataset describing the clinical and functional characteristics of a representative PSP cohort to allow researchers to investigate important unanswered questions in PSP.

Study population 50 patients with possible or probable PSP, according to established international criteria (i.e., MDS-PSP criteria); diagnosis confirmed by consensus review of a videotaped neurological examination by two neurologists with deep expertise in movement disorders. In addition, we will include 50 age and gender matched healthy controls.

Main study parameters/endpoints The primary study endpoints are the annual changes in the newly developed digital measurements, extracted from the Verily Study Watch. Secondary endpoints include standardized evaluations for motor, cognition, neuropsychological, quality of life and ADL assessments. Additionally, whole blood for DNA and serum will be collected in the PSP subjects, to use for e.g. genotyping and phenotyping.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness For data collection, the study assessor will visit each participant at home twice within an interval of 1 year ± 60 days. All study assessments are routine exams done in standard clinical practice and are generally well tolerated, which takes up to 2 hours each time. PSP subjects will also be asked to consent to a blood draw once. During their 1-year participation, each participant will wear the Verily Study Watch daily for up to 23 hours. This small, unobtrusive electronic device is easily worn and poses no significant safety risk. All participants will be asked to complete a set scheduled tasks twice a day, once a week, which altogether takes 15-20 minutes of their time.

As data collection is not performed for immediate diagnostic or therapeutic purposes, there will be no direct benefits for the subjects enrolled in this study. Patients may indirectly benefit from the study, as their data contribute to providing novel etiological insights for improving the use of existing treatments, developing of new therapeutic approaches, and increasing the precision of personalized disease management.

ELIGIBILITY:
Inclusion Criteria (PSP cohort):

* Subject has possible or probable PSP, according to the established international criteria defined by the Movement Disorders Society (MDS-PSP criteria, Höglinger et al, 2017); diagnosis is confirmed based on by consensus review process. In addition to the diagnosis of the own treating neurologist, the diagnosis always needs to be confirmed by at least one neurologist with deep expertise in movement disorders. The videotaped neurological examination as obtained during visit 1 will be used by the expert neurologist.
* Subject is an adult, at least 50 years of age.
* Subject can read and understand Dutch.
* Subject has completed the Informed Consent, as approved by the Institutional Review Board (IRB).
* Subject is willing, competent, and able to comply with all aspects of the protocol.
* Subject is able to walk at least 5 steps with or without minimal assistance (ie, stabilization of 1 arm or use of a cane or walker).

Inclusion Criteria (HC cohort):

* Subject has no neurological or musculoskeletal disorder or any other condition that impairs movement, gait, or balance, in the opinion of the Investigator.
* Subject is an adult, at least 50 years of age.
* Subject can read and understand Dutch.
* Subject has completed the Informed Consent, as approved by the IRB.
* Subject is willing, competent, and able to comply with all aspects of the protocol.
* Subject is able to walk at least 5 steps with or without minimal assistance (i.e., stabilization of 1 arm or use of a cane or walker).

Exclusion Criteria (PSP and HC cohorts):

* Subject has an additional condition or situation that, in the opinion of the Investigator, makes the subject inappropriate for participation in the study.
* For Study Watch: subject is allergic to nickel.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: PSP-cohort: any adult with PSP who meets the inclusion criteria and does not meet the exclusion criteria.
  HC-cohort: any adult who meets the inclusion criteria and does not meet the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2024-08-14 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
Annual change in digital biomarkers for gait | From baseline till one year follow-up
  Identify (a combined set of) gait-related features extracted from wearable sensor data, that are relevant for patients and that are sensitive to disease progression in PSP patients. Which outcome and which Unit of Measure for gait will be selected cannot be defined on forehand, as this is part of the analytical approach.
Annual change in digital biomarkers for bradykinesia | From baseline till one year follow-up
  Identify (a combined set of) bradykinesia-related features extracted from wearable sensor data, that are relevant for patients and that are sensitive to disease progression in PSP patients. Which outcome and which Unit of Measure for bradykinesia will be selected cannot be defined on forehand, as this is part of the analytical approach.
Annual change in digital biomarkers for falls | From baseline till one year follow-up
  Identify (a combined set of) falls-related features extracted from wearable sensor data, that are relevant for patients and that are sensitive to disease progression in PSP patients. Which outcome and which Unit of Measure for falls will be selected cannot be defined on forehand, as this is part of the analytical approach.
Annual change in digital biomarkers for rising from a chair | From baseline till one year follow-up
  Identify (a combined set of) features related to rising from a chair extracted from wearable sensor data, that are relevant for patients and that are sensitive to disease progression in PSP patients. Which outcome and which Unit of Measure for rising from a chair will be selected cannot be defined on forehand, as this is part of the analytical approach.

SECONDARY OUTCOMES:
Annual change in digital biomarker for motor performance | Baseline till one year follow-up
  Standardized evaluation, by means of 8 tasks, included in the Virtual Motor Examination. Which outcome and which Unit of Measure for motor performance will be selected cannot be defined on forehand, as this is part of the analytical approach.
Annual change in cognition | Baseline till one year follow-up
  Cognition will be assessed by means of the Mini-Mental State Examination version 2 (MMSE-2), on a 0-30-point scale.
Annual change in D-KEFS trail making test | Baseline till one year follow-up
  D-KEFS (Delis-Kaplan Executive Function System) trail making test is a neuropsychological test for executive functioning, with scores in seconds to perform the task.
Annual change in semantic fluency | Baseline till one year follow-up
  The semantic fluency test is a neuropsychological assessment, measuring executive function and semantic memory. The score entails the number of correct and unique words produced within a 60 seconds timeframe.
Annual change in quality of life | Baseline till one year follow-up
  Quality of life is captured by means of a general scale, i.e., EQ-5D-5L. The EQ-5D-5L consists of 2 parts: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement.
Annual change in Activities of Daily Living (ADL) performance | Baseline till one year follow-up
  Modified Schwab & England Activities of Daily Living is a method of assessing the capabilities of people with impaired mobility. The scale uses percentages to represent how much effort and dependence on others people need to complete daily chores.

CONTACTS AND LOCATIONS:
Overall Officials: Bastiaan R Bloem, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Medical Center, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The dataset generated in this study will become available to qualified researchers worldwide, provided research questions are approved by the Research and Data Sharing Review Committee (RDSRC). The RDSRC will protect subjects' privacy by limiting the availability of the study data and controlling access to sources of information that might potentially be used to identify the individual subjects associated with the bio-specimen analysis. The RDSRC will assess the relevance and scientific quality of research proposals for which study data or material is requested. These responsibilities include the consideration of applications for:
  * access to the resources obtained in this study, including data or biomaterials
  * applications for endorsement of a scientific project using study materials;
  * applications for endorsement of a clinical study using study materials.
Supporting Information: Study Protocol
Time Frame: Not decided yet.
Access Criteria: No list of criteria is available yet.